CLINICAL TRIAL: NCT02045563
Title: Genetic Polymorphisms, Hepatic Steatosis and Lipid Anomalies in Diabetic Patients
Brief Title: Genetic Polymorphisms, Steatosis and Diabetes
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PETIT PARI 2011
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Type 1 and 2 Diabetes
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Patients with type-1 diabetes
  Interventions: Other: prise de sang; Other: magnetic resonance imaging and magnetic resonance spectroscopy
- Patients with type-2 diabetes
  Interventions: Other: prise de sang; Other: magnetic resonance imaging and magnetic resonance spectroscopy
- Volontaires sains
  Interventions: Other: prise de sang; Other: magnetic resonance imaging and magnetic resonance spectroscopy

INTERVENTIONS:
Other: prise de sang
Other: magnetic resonance imaging and magnetic resonance spectroscopy

SUMMARY:
* Our research hypothesis is to show that a certain number of genetic polymorphisms of the proteins involved in glucose, lipid and adipocyte metabolism are factors that favour the development of steatosis in patients with Type 2 diabetes.
* We also wish to evaluate more thoroughly lipid anomalies associated with the presence of steatosis, notably with regard to monocyte expression of LDL receptors. We hypothesize that hepatic steatosis is accompanied by activation of transcription factors involved in lipogenesis, notably SREBP factors. The activation of these factors could cause an increase in the expression of LDL receptors, leading to increased LDL catabolism.
* Chronological description of the study During an outpatient consultation at the endocrinology department, diabetic patients, programmed to undergo an examination to assess their diabetes will be invited to participate in the study. Once written informed consent has been provided and clinical data has been recorded, patients with type 1 or type 2 diabetes will have standard biological examination, which is systematically done in such patients (Fasting glycemia, HBA1c, aspartate aminotransferase, alanine amino transferase, Gammaglutamyl-transferases, PAL, bilirubin, blood proteins, albuminemia, Total Cholesterol total, HDL cholesterol, triglycerides, Sedimentation Rate, C-reactive protein, fibrinogen).

As well as the systematic biological tests, 3 additional tubes will be taken to screen for genetic polymorphism in 3 proteins (Microsomal Transfer Protein, Adiponectin receptor - 1, Apolipoprotein A - II).

IN addition, magnetic resonance imaging and magnetic resonance spectroscopy will be done to look for the presence of liver steatosis and to measure carotid intima-media thickness.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria Type-2 diabetics:

* Type 2 diabetes
* HbA1C>6.5%
* 27<BMI<55

Inclusion criteria Type-1 diabetics:

* Type 1 diabetes
* BMI<55 Diagnosis of type-1 diabetes based on the clinical history of the patient and/or the presence of anti-glutamate decarboxylase auto antibodies and/or a plasma level of C peptide below 0,5 ng/l.

Inclusion criteria healthy volunteers:

* Non diabetic
* Alcohol consumption < 2 glasses per day
* Without hyperglycemic treatment (corticoids, ...)
* Without liver disease (cirrhosis, hepatitis, ...)

Exclusion Criteria:

* Pacemaker
* Daily alcohol consumption above 4 glasses per day
* Patients treated with Glitazones during the 3 months preceding inclusion
* Presence of implants
* Claustrophobia
* Patient < 18 years
* Patient under guardianship or not intellectually independent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of type 2 diabetes over 18 subjects treated with diet alone or with oral antidiabetic glitazones outside of patients with type 1 and of age-matched healthy volunteers and sex.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2007-10-15 (Actual); Primary Completion 2015-03-25 (Actual); Study Completion 2015-03-25 (Actual)

PRIMARY OUTCOMES:
Determination of the existence of liver steatosis measured by magnetic resonance spectroscopy spectrometry | At inclusion

SECONDARY OUTCOMES:
Measurement of monocyte expression of LDL receptors | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France